CLINICAL TRIAL: NCT00818623
Title: An Open-Label, Multi-Center, Parallel and Sequential, Ascending Single Dose Study Investigating the Pharmacokinetics, Pharmacodynamics and Safety of FE200486 in Prostate Cancer Patients
Brief Title: Investigation of a New Trial Drug (FE200486) in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS07
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2009-03-31 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2011-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Degarelix 120 mg (20 mg/mL) (Experimental): Degarelix 120 mg (20 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 120 mg (40 mg/mL) (Experimental): Degarelix 120 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 160 mg (40 mg/mL) (Experimental): Degarelix 160 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 200 mg (40 mg/mL) (Experimental): Degarelix 200 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 200 mg (60 mg/mL) (Experimental): Degarelix 200 mg (60 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 240 mg (40 mg/mL) (Experimental): Degarelix 240 mg (40 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 240 mg (60 mg/mL) (Experimental): Degarelix 240 mg (60 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 320 mg (60 mg/mL) (Experimental): Degarelix 320 mg (60 mg/mL)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Degarelix (120 mg (20 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 120 mg (20 mg/mL)
Drug: Degarelix — Degarelix (120 mg (40 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 120 mg (40 mg/mL)
Drug: Degarelix — Degarelix (160 mg (40 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 160 mg (40 mg/mL)
Drug: Degarelix — Degarelix (200 mg (40 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 200 mg (40 mg/mL)
Drug: Degarelix — Degarelix (200 mg (60 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 200 mg (60 mg/mL)
Drug: Degarelix — Degarelix (240 mg (40 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 240 mg (40 mg/mL)
Drug: Degarelix — Degarelix (240 mg (60 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 240 mg (60 mg/mL)
Drug: Degarelix — Degarelix (320 mg (60 mg/mL)) was given as a subcutaneous injection
  Other Names: FE200486
  Arms: Degarelix 320 mg (60 mg/mL)

SUMMARY:
The purpose of this trial was to find an optimal dose for a new trial drug - degarelix (FE200486) - in the treatment of prostate cancer. Furthermore the safety of the drug was studied. Patients participating were treated with FE200486 on one occasion. Thereafter they came in for visits following a specific schedule until blood samples showed that there was no further effect.

DETAILED DESCRIPTION:
Degarelix was not FDA regulated at the time of the trial. After completion of the trial degarelix has been approved by the FDA and is thus an FDA regulated intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any trial related procedures
* Male patient with proven prostate cancer in need for endocrine treatment, except for neoadjuvant hormonal therapy
* ECOG score to be equal to or above 2
* Testosterone level within age-specific normal range
* PSA value equal to or above 2 ng/ml
* Life expectancy of at least 6 months

Exclusion Criteria:

* Previous or current hormonal treatment of prostate cancer
* Recent or current treatment with any drugs modifying the testosterone level
* Candidate for curative treatment such as prostatectomy or radiotherapy
* History of severe asthma, anaphylactic reactions or Quincke's Oedema
* Hypersensitivity towards any component of FE200486
* Cancer disease within the last ten years except for prostate cancer and some skin cancers
* Signs of liver impairment shown as elevated serum ALT or serum bilirubin
* Other laboratory abnormalities that judged by the investigator would interfere with the patients participation in the trial or the evaluation of the trial results
* Presenting with significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, haematological, dermatological or infectious disorder. In addition any other condition such as excessive alcohol or drug abuse that may interfere with trial participation or influence the conclusion of the trial as judged by the investigator
* Mental incapacity or language barrier
* Having received an investigational product within the last 12 weeks preceding the trial
* Previous participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2002-11; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (30):
- Denmark (3):
  - Rigshospitalet, Copenhagen
  - KAS Glostrup, Glostrup Municipality
  - KAS Herlev, Herlev
- Finland (6):
  - Marian Sairaala, Helsinki
  - P-K Keskussairaala, Joensuu
  - Vuorikadun lääkäriasema, Kuopio
  - OYS, Oulu
  - Kirugikeskus, Seinäjoki
  - TAYS, Tampere
- Hungary (6):
  - Bajcsy-Zsilinszky Hospital, Urology, Budapest
  - Jahn Ferenc Dél Pesti Hospital, Urology, Budapest
  - Péterfy Hospital, Urology, Budapest
  - Bács-Kiskun County Hospital, Urology, Kecskemét
  - Hospital of Local Gov. Szeged, Urology, Szeged
  - MÁV Hospital, Urology, Szolnok
- Sentralsykehuset i Rogland, Stavanger, Norway
- Romania (4):
  - CF2 Hospital - Bucharest, Urology, Bucharest
  - Dr. Th Burghele Hospital, Bucharest
  - Fundeni Hospital - Bucharest, Urology, Bucharest
  - County Hospital - Timisoara, Urology, Timișoara
- Russia (5):
  - City Hospital #1, State Med Univ/Urology, Moscow
  - Institute of Urology of MoH, Moscow
  - Moscow City Hospital #60, Urology, Moscow
  - City Hospital #15, Urology Department, Saint Petersburg
  - City Hospital #26, Urology Department, Saint Petersburg
- Sweden (5):
  - Sahlgrenska Universitetssjukehuset, Gothenburg
  - Helsingborgs Lasaret, Helsingborg
  - Universitetssjukehuset, MAS, Malmo
  - University Hospital, Örebro, Örebro
  - Akademiska Sjukhuset Uppsala, Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- Degarelix 120mg (20mg/mL): Degarelix 120 mg (20 mg/mL)
- Degarelix 120mg (40mg/mL): Degarelix 120 mg (40 mg/mL)
- Degarelix 160mg (40mg/mL): Degarelix 160 mg (40 mg/mL)
- Degarelix 200mg (40mg/mL): Degarelix 200 mg (40 mg/mL)
- Degarelix 200mg (60mg/mL): Degarelix 200 mg (60 mg/mL)
- Degarelix 240mg (40mg/mL): Degarelix 240 mg (40 mg/mL)
- Degarelix 240mg (60mg/mL): Degarelix 240 mg (60 mg/mL)
- Degarelix 320mg (60mg/mL): Degarelix 320 mg (60 mg/mL)
Period: Overall Study
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Started | 26 | 12 | 13 | 24 | 27 | 24 | 27 | 27
Intent-to-treat (ITT) Population | 25 (One participant in this group was randomized but never received any treatment.) | 12 | 12 (One participant in this group was randomized but never received any treatment.) | 24 | 24 (Three participants in this group were randomized but never received any treatment.) | 24 | 24 (Three participants in this group were randomized but never received any treatment.) | 27
Completed | 24 | 8 | 9 | 19 | 23 | 21 | 23 | 26
Not Completed | 2 | 4 | 4 | 5 | 4 | 3 | 4 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Bad prostate specific antigen response | 0 | 3 | 2 | 5 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Need of additional treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of trial drug at site | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL) | Total
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 0 | 2 | 2 | 4 | 2 | 6 | 6 | 29
  >=65 years | 18 | 12 | 10 | 22 | 20 | 22 | 18 | 21 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (10.3) | 73.8 (3.97) | 70.1 (8.08) | 74.3 (6.48) | 71.5 (8.27) | 73.1 (5.96) | 71.7 (9.54) | 71.1 (6.87) | 71.9 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 27 | 172
Curative intent [Number; unit: participants] — A curative intent of Yes refers to participants who have been castrated via radical prostatectomy or radiotherapy.
  participants
    Yes | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 1 | 7
    No | 25 | 12 | 10 | 21 | 23 | 24 | 24 | 26 | 165
Gleason score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    0-1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    2-4 | 4 | 0 | 2 | 1 | 5 | 2 | 5 | 12 | 31
    5-6 | 4 | 7 | 5 | 6 | 3 | 6 | 6 | 6 | 43
    7-10 | 17 | 5 | 5 | 17 | 16 | 16 | 13 | 9 | 98
Stage of prostate cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 10 | 1 | 3 | 3 | 1 | 6 | 8 | 14 | 46
    Locally advanced | 6 | 6 | 5 | 14 | 8 | 10 | 5 | 9 | 63
    Metastatic | 9 | 3 | 4 | 6 | 12 | 6 | 10 | 2 | 52
    Not classifiable | 0 | 2 | 0 | 1 | 3 | 2 | 1 | 2 | 11
Body mass index [Mean (Standard Deviation); unit: kilgram per square meter] | 26.2 (2.97) | 26.6 (4.58) | 26.3 (3.74) | 25.9 (2.99) | 24.5 (2.92) | 26.9 (3.18) | 24.8 (2.72) | 27.1 (3.63) | 26.0 (3.32)
Serum prostate-specific antigen levels [Median (Full Range); unit: nanogram per milliliter] | 42.5 [3.0 to 4509] | 58.8 [9.7 to 5514] | 109 [4.1 to 1079] | 32.3 [3.8 to 1474] | 46.9 [2.3 to 6450] | 31.0 [4.5 to 357] | 31.9 [5.2 to 3490] | 23.8 [1.7 to 731] | 37.9 [1.7 to 6450]
Serum testosterone levels [Median (Full Range); unit: nanogram per milliliter] | 4.30 [2.37 to 12.5] | 3.10 [1.08 to 6.91] | 3.02 [1.65 to 5.12] | 4.64 [1.97 to 7.93] | 5.60 [3.01 to 9.36] | 4.02 [1.49 to 12.5] | 4.46 [1.81 to 11.2] | 3.68 [1.45 to 7.26] | 4.16 [1.08 to 12.5]
Time since prostate cancer diagnosis [Mean (Standard Deviation); unit: days] | 83.2 (157) | 65.9 (53.5) | 222 (328) | 146 (298) | 252 (560) | 313 (837) | 121 (425) | 46.6 (54.4) | 156 (439)
Weight [Mean (Standard Deviation); unit: kilogram] | 77.8 (12.4) | 82.2 (12.1) | 80.7 (11.8) | 78.2 (13.7) | 74.2 (9.88) | 81.5 (10.7) | 73.5 (9.55) | 81.7 (11.1) | 78.4 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Time From Dosing Until Testosterone Levels >0.5 ng/mL
Description: Intent-to-treat (ITT) population. This outcome measure is based on one testosterone value >0.5 ng/mL at Day 28 onwards.
Time Frame: 3 months
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
days | 84 [63 to 119] | 63 [28 to 133] | 70 [28 to 98] | 140 [112 to 147] | 84 [35 to 112] | 140 [112 to 182] | 87.5 [28 to 140] | 133 [91 to 154]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.0000586, Log Rank

2. Secondary Outcome: Number of Participants With Testosterone Level ≤0.5 ng/mL for at Least 28 Days
Description: The table shows the number of participants with testosterone level ≤0.5 ng/mL for at least 28 days.
Time Frame: Two - six months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
participants | 21 [66.1 to 95.8] | 8 [33.7 to 86.0] | 6 [22.9 to 78.0] | 24 [85.8 to 100] | 18 [52.6 to 87.9] | 22 [72.9 to 99.4] | 15 [40.3 to 78.4] | 24 [69.4 to 96.3]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.0014, Kruskal-Wallis
Statistical Analysis 2: Comparison: Degarelix 120mg (20mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 87.5, 95% CI [66.1 to 95.8]
Statistical Analysis 3: Comparison: Degarelix 120mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 66.7, 95% CI [33.7 to 86]
Statistical Analysis 4: Comparison: Degarelix 160mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 54.5, 95% CI [22.9 to 78]
Statistical Analysis 5: Comparison: Degarelix 200mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 100, 95% CI [85.8 to 100]
Statistical Analysis 6: Comparison: Degarelix 200mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 75, 95% CI [52.6 to 87.9]
Statistical Analysis 7: Comparison: Degarelix 240mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 95.7, 95% CI [72.9 to 99.4]
Statistical Analysis 8: Comparison: Degarelix 240mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 62.5, 95% CI [40.3 to 78.4]
Statistical Analysis 9: Comparison: Degarelix 320mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 28 days; Test type: Superiority or Other; Percentage of participants castrated = 88.9, 95% CI [69.4 to 96.3]

3. Secondary Outcome: Number of Participants With Testosterone Level ≤0.5 ng/mL for at Least 84 Days
Description: The table shows the number of participants with testosterone level ≤0.5 ng/mL for at least 84 days.
Time Frame: 3 months
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
participants | 11 [25.6 to 64] | 4 [12.1 to 64.3] | 3 [8.3 to 60.6] | 20 [61.5 to 93.4] | 11 [28.3 to 67.4] | 18 [58.8 to 92.8] | 12 [29.1 to 67.8] | 19 [49.4 to 83.9]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.0031, Kruskal-Wallis
Statistical Analysis 2: Comparison: Degarelix 120mg (20mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 45.8, 95% CI [25.6 to 64]
Statistical Analysis 3: Comparison: Degarelix 120mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 38.1, 95% CI [12.1 to 64.3]
Statistical Analysis 4: Comparison: Degarelix 160mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 32.7, 95% CI [8.3 to 60.6]
Statistical Analysis 5: Comparison: Degarelix 200mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 83.3, 95% CI [61.5 to 93.4]
Statistical Analysis 6: Comparison: Degarelix 200mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 49.4, 95% CI [28.3 to 67.4]
Statistical Analysis 7: Comparison: Degarelix 240mg (40mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 82, 95% CI [58.8 to 92.8]
Statistical Analysis 8: Comparison: Degarelix 240mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 50, 95% CI [29.1 to 67.8]
Statistical Analysis 9: Comparison: Degarelix 320mg (60mg/mL); Percentage of participants castrated (testosterone ≤0.5 ng/mL) for at least 84 days; Test type: Superiority or Other; Percentage of participants castrated = 70.4, 95% CI [49.4 to 83.9]

4. Secondary Outcome: Time to Testosterone Castration (Testosterone ≤0.5 ng/mL)
Description: Time to testosterone castration was calculated as the number of days from dosing to the first scheduled visit when testosterone was less than 0.5 ng/mL.
Time Frame: 3 months
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
days | 1 [1 to 7] | 1 [1 to 3] | 1.5 [1 to 2] | 1.5 [1 to 7] | 2 [1 to 14] | 1.5 [1 to 7] | 2 [1 to 3] | 1 [1 to 3]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.0866, Log Rank

5. Secondary Outcome: Time to 50% Reduction in Prostate-specific Antigen Levels
Description: The time to 50% prostate-specific antigen (PSA) reduction from baseline was defined as the number of days from dosing to the first visit where a 50% reduction in PSA level was reached.
Time Frame: 3 months
Population: ITT population. Patients who did not achieve the actual level of reduction were censored as of the time from dosing for the last available observation.
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
days | 14 [7 to 28] | 21 [7 to 21] | 14 [7 to 28] | 14 [7 to 35] | 14 [7 to 49] | 14 [7 to 35] | 14 [7 to 35] | 14 [7 to 35]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.033, Log Rank

6. Secondary Outcome: Time to 90% Reduction in Prostate-specific Antigen Levels
Description: The time to 90% prostate-specific antigen (PSA) reduction from baseline was defined as the number of days from dosing to the first visit where a 90% reduction in PSA level was reached.
Time Frame: 3 months
Population: ITT population. Participants who did not achieve the actual level of reduction were censored as of the time from dosing for the last available observation.
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
days | 31.5 [14 to 56] | 35 [21 to 91] | 42 [28 to 70] | 35 [14 to 98] | 28 [14 to 63] | 42 [21 to 112] | 35 [14 to 77] | 45.5 [21 to 112]
Statistical Analysis 1: Comparison: Degarelix 120mg (20mg/mL) vs Degarelix 120mg (40mg/mL) vs Degarelix 160mg (40mg/mL) vs Degarelix 200mg (40mg/mL) vs Degarelix 200mg (60mg/mL) vs Degarelix 240mg (40mg/mL) vs Degarelix 240mg (60mg/mL) vs Degarelix 320mg (60mg/mL); Test type: Superiority or Other; p = 0.131, Log Rank

7. Secondary Outcome: Evaluation of Liver Function Tests
Description: The figures presents the number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferase levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
participants
  Abnormal alanine aminotransferase (ALAT) | 9 | 2 | 3 | 7 | 8 | 4 | 6 | 6
  Abnormal aspartate aminotransferase | 6 | 3 | 1 | 4 | 7 | 3 | 5 | 5
  Abnormal bilirubin | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1
  ALAT >3x ULN | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Participants With Markedly Abnormal Change in Vital Signs and Body Weight
Description: Vital signs and body weight included incidence of markedly abnormal changes in blood pressure (systolic and diastolic), pulse, and body weight at the end of trial as compared to baseline. The table presents the number of participants in each group with normal baseline and markedly abnormal value post-baseline.
Time Frame: 3 months
Population: ITT population. The first value in the category represents the actual clinical reading and the second is the change from baseline for blood pressure (units: millimeters of mercury) and heart rate (units:beats per minute). The weight category includes participants whose percent weight change from baseline fit the stated ranges.
Measure: Number; unit: participants
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Number analyzed (Participants) | 25 | 12 | 12 | 24 | 24 | 24 | 24 | 24
participants
  Diastolic blood pressure <=50 and decrease >=15 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Diastolic blood pressure >=105 and increase >=15 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Systolic blood pressure <=90 and decrease >=20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure >=180 and increase >=20 | 0 | 0 | 1 | 3 | 1 | 2 | 1 | 2
  Heart rate <=50 and decrease >=15 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Heart rate >=120 and increase >=15 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Body weight decrease of >=7 percent | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Body weight increase of >=7 percent | 2 | 1 | 1 | 2 | 1 | 0 | 3 | 1

ADVERSE EVENTS:
Arm/Group | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Serious Adverse Events (participants affected / at risk) | 2 | 2 | 1 | 2 | 1 | 4 | 3 | 4
Other Adverse Events (participants affected / at risk) | 14 | 10 | 7 | 20 | 14 | 22 | 10 | 19
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Cardiac failure (Cardiac disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Acute myocardial infarction (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Angina pectoris (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Myocardial infarction (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Vomiting (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Condition aggravated (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Oedema (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Gangrene (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Pneumonia (Infections and infestations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Gamma-glutamyltransferase increased (Investigations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Inervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Areflexia (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Ischaemic stroke (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Paraplegia (Nervous system disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Spinal cord compression (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Completed suicide (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Depression (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Haematuria (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Amputation revision (Surgical and medical procedures) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Deep vein thrombosis (Vascular disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Hypertension (Vascular disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 120mg (20mg/mL) | Degarelix 120mg (40mg/mL) | Degarelix 160mg (40mg/mL) | Degarelix 200mg (40mg/mL) | Degarelix 200mg (60mg/mL) | Degarelix 240mg (40mg/mL) | Degarelix 240mg (60mg/mL) | Degarelix 320mg (60mg/mL)
Angina pectoris (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 2/27 (2)
Atrial fibrillation (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Bradycardia (Cardiac disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Cataract (Eye disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Glaucoma (Eye disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Diarrhoea (Gastrointestinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 3/24 (3) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 1/27 (1)
Nausea (Gastrointestinal disorders) | 0/25 (0) | 2/12 (2) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Dyspepsia (Gastrointestinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Anal fissure (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Stomach discomfort (Gastrointestinal disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site pain (General disorders) | 1/25 (1) | 2/12 (2) | 1/12 (1) | 2/24 (2) | 1/24 (1) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Injection site erythema (General disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 3/24 (3) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Fatigue (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (3) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Chest pain (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Chills (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/27 (0)
Feeling of body temperature change (General disorders) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site induration (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site pruritus (General disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Oedema peripheral (General disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (2) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Injection site swelling (General disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Urinary tract infection (Infections and infestations) | 3/25 (3) | 0/12 (0) | 0/12 (0) | 1/24 (1) | 0/24 (0) | 3/24 (3) | 2/24 (2) | 2/27 (2)
Nasopharyngitis (Infections and infestations) | 1/25 (1) | 2/12 (2) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 1/27 (1)
Cystitis (Infections and infestations) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Oral fungal infection (Infections and infestations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Blood alkaline phosphatase increased (Investigations) | 3/25 (3) | 0/12 (0) | 0/12 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Gamma-glutamyltransferase increased (Investigations) | 3/25 (3) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (3) | 0/24 (0) | 0/27 (0)
Alanine aminotransferase increased (Investigations) | 4/25 (4) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Aspartate aminotransferase increased (Investigations) | 2/25 (2) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Blood pressure increased (Investigations) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 2/27 (3)
Hepatic enzyme increased (Investigations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Prostatic specific antigen increased (Investigations) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 1/12 (2) | 0/12 (0) | 1/24 (1) | 3/24 (3) | 1/24 (1) | 1/24 (1) | 1/27 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 1/12 (1) | 1/24 (1) | 0/24 (0) | 1/24 (2) | 1/24 (1) | 0/27 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1/25 (1) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/27 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Headache (Nervous system disorders) | 0/25 (0) | 2/12 (2) | 0/12 (0) | 3/24 (3) | 0/24 (0) | 3/24 (3) | 0/24 (0) | 0/27 (0)
Dizziness (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2) | 0/27 (0)
Hypoaesthesia (Nervous system disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Insomnia (Psychiatric disorders) | 2/25 (2) | 0/12 (0) | 1/12 (1) | 2/24 (2) | 1/24 (1) | 0/24 (0) | 1/24 (2) | 0/27 (0)
Nervousness (Psychiatric disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nightmare (Psychiatric disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nocturia (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 0/12 (0) | 3/24 (3) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Haematuria (Renal and urinary disorders) | 0/25 (0) | 0/12 (0) | 1/12 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/27 (0)
Prostatitis (Reproductive system and breast disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 1/27 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 0/12 (0) | 0/12 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/25 (1) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6/25 (6) | 2/12 (2) | 0/12 (0) | 5/24 (6) | 5/24 (5) | 5/24 (5) | 2/24 (2) | 1/27 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0/25 (0) | 1/12 (2) | 0/12 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0) | 0/27 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0/25 (0) | 0/12 (0) | 1/12 (1) | 1/24 (2) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Hot flush (Vascular disorders) | 4/25 (4) | 1/12 (1) | 3/12 (4) | 12/24 (12) | 6/24 (6) | 9/24 (9) | 4/24 (4) | 9/27 (9)
Flushing (Vascular disorders) | 0/25 (0) | 1/12 (1) | 0/12 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.